CLINICAL TRIAL: NCT01250457
Title: Topical Timolol for the Treatment of Benign Vascular Periocular Lesions
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unknown, PI has left the institution. There was no enrollment.
Sponsor: Loyola University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202688
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Benign Vascular Periocular Lesions
MeSH Terms: interventions — Timolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Topical timolol (Experimental): topical Timolol 0.5% solution applied twice daily
  Interventions: Drug: topical Timolol

INTERVENTIONS:
Drug: topical Timolol — topical Timolol 0.5% solution applied twice daily
  Other Names: Timoptic

SUMMARY:
The purpose of this research is to find out if the use of topical timolol 0.5% solution applied twice daily will help to shrink rosacea lesions around the eye.

DETAILED DESCRIPTION:
Benign vascular tumors of the eyelid are common causes of ocular morbidity. Capillary hemangiomas in children cause refractive and occlusive amblyopia. In adults, Rosacea-associated eyelid telangiectasis and sclerosis can result in keratitis and corneal neovascularization. Corticosteroid therapy of benign vascular lesions risks sight-threatening complications including central retinal artery occlusion and significant systemic morbidity. Alternatively, oral and intravenous beta-blockers have been reported to induce regression of benign vascular lesions. One recent report documented efficacy of topical timolol in treating a large capillary hemangioma of the eyelid in a child. Topical application reduces systemic side effects of beta-blockers including bradycardia, hypotension, heart block, and bronchospasm. This one-year prospective case-control series will investigate whether topical Timolol 0.5% solution applied twice daily causes significant regression of benign vascular periocular lesions.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a benign vascular periocular lesion

Exclusion Criteria:

* Allergy to timolol or beta-blocker class of drugs
* Lesion characteristics concerning for atypia or malignancy including madarosis, ulceration, and recurrence after previous surgery.
* Intraocular Pressure less than 10 mm Hg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
lesion resolution | 1 year
  Pre-treatment and post-treatment lesion size will then be compared to determine whether twice-daily topical application of timolol 0.5% solution alters the morphometry of benign vascular periocular lesions.

CONTACTS AND LOCATIONS:
Overall Officials: David Yoo, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States